CLINICAL TRIAL: NCT05321394
Title: Adaptive, Randomized, Non-inferiority Trial on the Use of Monoclonal Antibodies or Antivirals in Outpatients With Mild or Moderate COVID-19
Brief Title: Non-inferiority Trial on Treatments in Early COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government); Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Evelina Tacconelli, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MANTICO 2; 2021-002612-31 (EudraCT Number)
Record Dates: First submitted 2022-04-07; First posted 2022-04-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: COVID-19
Keywords: Coronavirus Infections; Monoclonal antibodies; Sotrovimab; Tixagevimab Cilgavimab; Nirmatrelvir Ritonavir
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — sotrovimab; cilgavimab and tixagevimab drug combination; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sotrovimab (Active Comparator): Sotrovimab 500 mg administered in 100 mL prefilled 0.9% sodium chloride injection infusion solution over 1/2 hour
  Interventions: Drug: Sotrovimab
- Tixagevimab Cilgavimab (Experimental): 300 mg of tixagevimab and 300 mg of cilgavimab administered as two separate consecutive intramuscular injections
  Interventions: Drug: Tixagevimab Cilgavimab
- Nirmatrelvir Ritonavir (Experimental): 300 mg nirmatrelvir (two 150 mg tablets) with 100 mg ritonavir (one 100 mg tablet) with all three tablets taken together twice daily for 5 days
  Interventions: Drug: Nirmatrelvir Ritonavir

INTERVENTIONS:
Drug: Sotrovimab — Single intravenous infusion of sotrovimab 500 mg (500 mg/8 mL), administered in 100 mL prefilled 0.9% sodium chloride injection infusion solution over 1/2 hour.
  Arms: Sotrovimab
Drug: Tixagevimab Cilgavimab — 2 subsequent injections:
  1. tixagevimab 300mg/3mL (100mg/mL)
  2. cilgavimab 300mg/3mL (100mg/mL)
  Arms: Tixagevimab Cilgavimab
Drug: Nirmatrelvir Ritonavir — 300 mg nirmatrelvir (two 150 mg tablets) with 100 mg ritonavir (one 100 mg tablet) with all three tablets taken together twice daily for 5 days
  Arms: Nirmatrelvir Ritonavir

SUMMARY:
The study aims at assessing the non-inferiority of tixagevimab plus cilgavimab and nirmatrelvir plus ritornavir vs. sotrovimab (reference standard due to the wider evidence gathered on its efficacy) on COVID-19 progression in a real-life setting of outpatients aged at least 50 years at an early stage of the disease. The progression of COVID-19 disease (hospitalization, need for supplementary oxygen therapy at home, death) within 14 days of randomisation is the composite outcome variable on which the calculation of the sample size is based. Based on available data regarding the reduction in the number of hospitalisations and medical visits with the use of sotrovimab at an early-stage of COVID-19, a disease progression of 1% has been estimated in the reference arm. 3% delta margin was considered clinically relevant, taking into account both the estimates of disease progression in the study population in absence of early treatment (7%, based on national data) and the efficacy of the reference standard. Therefore, 1095 participants will be randomly assigned in an equal ratio between the reference standard and each of the other two experimental arms (1:1:1). Randomization will be computer-generated in permuted blocks with a stratification based on site.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Informed consent by the subject or legally authorized representative
* Laboratory-confirmed SARS-CoV-2 infection, as determined by PCR or other commercial or public health assay in any specimen, no more than 4 days prior to the study drug administration
* Peripheral oxygen saturation ≥ 94% on room air and not requiring supplemental oxygen
* Onset of symptom is no more than 4 days prior to the study drug administration. Onset time of symptom is defined as the time when the patient experienced the presence of at least one of the following (but not limited to) SARS-CoV-2 infection-associated symptom (FDA, September 2020): nasal obstruction or congestion, cough, fever > 37.3 °C, sore throat, body pain or muscle pain, headache, loss of taste or smell, nausea or vomiting, diarrhoea

Exclusion Criteria:

* Previously or currently hospitalized or requiring hospitalization
* Respiratory distress with respiratory rate ≥ 25 breaths/min
* Heart rate ≥ 125 beats per minute
* Peripheral oxygen saturation ≤ 93% on room air at sea level
* Known allergies to any of the components used in the formulation of the interventions
* Severe renal impairment (eGFR <30 mL/min)
* Severe hepatic impairment (Child-Pugh Class C)
* Co-administration with drugs highly dependent on CYP3A for clearance and for which elevated concentrations are associated with serious and/or life-threatening reactions
* Co-administration with potent CYP3A inducers
* Hemodynamic instability requiring use of pressors within 24 hours of randomization
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that could potentially lead to hospitalization in within 30 days
* Any co-morbidity requiring surgery within 7 days or that is considered life-threatening within 90 days
* History of a positive SARS-CoV-2 test prior to the one serving as eligibility for this study
* Other investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing
* Previous treatment with a SARS-CoV-2 specific monoclonal antibody
* History of convalescent COVID-19 plasma treatment
* Participation, within the last 30 days, in a clinical study involving an investigational intervention
* Pregnancy or breast feeding
* Investigator site personnel directly affiliated with this study
* Sexually active women of childbearing potential or sexually active men who are unwilling to practice effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose
* Inability to participate to the study follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
COVID-19 progression | 14 days
  (1) hospitalization or (2) need of supplemental oxygen therapy at home or (3) death within 14 days of randomisation

SECONDARY OUTCOMES:
Visits to the Emergency Room | 28 days
  Number of visits to the Emergency Room without subsequent hospitalization within 28 days of randomization
Duration of supplemental oxygen therapy | 90 days
  Days of supplemental oxygen therapy within 90 days of randomization
Duration of hospitalization | 90 days
  Days of any hospitalization within 90 days of randomization
Non-invasive ventilation | 28 days
  Rate of patients undergoing non-invasive ventilation within 28 days of randomization
Duration of non-invasive ventilation | 90 days
  Days of non-invasive ventilation within 90 days of randomization
Mechanical ventilation | 28 days
  Rate of patients undergoing mechanical ventilation within 28 of randomization
Duration of mechanical ventilation | 90 days
  Days of mechanical ventilation within 90 days of randomization
28-day mortality | 28 days
  Death rate at 28 days of randomization
90-day mortality | 90 days
  Death rate at 90 days of randomization
Duration of symptoms | 90 days
  Days of symptoms within 90 days of randomization

CONTACTS AND LOCATIONS:
Locations (19):
- Italy (19):
  - RCCS Policlinico di S. Orsola, Bologna
  - PO SS Trinità di Cagliari, Cagliari
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele, Catania
  - PO Garibaldi Nesima, Catania
  - Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - Ospedale S. Maria Annunziata, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera dei Colli, presidio ospedaliero Cotugno, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - AOU Policlinico, Palermo
  - Azienda Ospedaliera S. Maria della Misericordia, Perugia
  - Università degli Studi di Pescara, Pescara
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Ospedale San Paolo ASL 2 Savonese, Savona
  - AOU Città della Salute e Scienza, Presidio Molinette, Torino
  - Azienda Sanitaria Universitaria Giuliano-Isontina (ASUGI), Trieste
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
  - Azienda Ospedaliera di Verona, Verona

REFERENCES:
- [Derived] Mazzotta V, Mazzaferri F, Lanini S, Mirandola M, Cozzi Lepri A, Vergori A, Savoldi A, Santoro A, Maccarrone G, Mastrorosa I, Simonetti O, Zottis F, Nicastri E, Rosini G, Rovigo L, Tavernaro L, Sarmati L, Tascini C, Girardi E, Cattelan AM, Antinori A, Tacconelli E; MANTICO2/MONET study group. Pooled analysis of the MANTICO2 and MONET randomized controlled trials comparing drug efficacy for early treatment of COVID-19 during Omicron waves. J Infect. 2024 Nov;89(5):106294. doi: 10.1016/j.jinf.2024.106294. Epub 2024 Sep 27. PMID 39343244